CLINICAL TRIAL: NCT05734560
Title: Delivery of D2C7-IT and 2141-V11 Combination Immunotherapy in Residual Disease for Adult Patients With Newly Diagnosed MGMT Unmethylated Glioblastoma and Perilymphatic Subcutaneous Injections of 2141-V11
Brief Title: D2C7-IT and 2141-V11 in Newly Diagnosed GBM Patients
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Darell Bigner (Other)
Collaborators: Rockefeller University (Other)
Responsible Party: Sponsor-Investigator, Darell Bigner, Sponsor-Investigator, Duke University
Organization: Duke University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Pro00110119
Record Dates: First submitted 2023-02-07; First posted 2023-02-21 (Actual); Last update posted 2025-10-06 (Actual); Status verified 2025-10

CONDITIONS: Newly Diagnosed MGMT Unmethylated Glioblastoma
Keywords: D2C7; D2C7-IT; 2141-V11; Pro00110119; GBM; Glioblastoma; convection-enhanced delivery; CED; MGMT unmethylated
MeSH Terms: conditions — Glioblastoma | interventions — D2C7-(scdsFv)-PE38KDEL

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- D2C7-IT + 2141-V11 (Experimental): Single D2C7-IT intratumoral infusion (6920 ng/mL in 36 mL) over 72 hours followed by single 2141-V11 infusion (5 dose levels) over 7 hours followed by an injection of 2141-V11 in the cervical perilymphatic subcutaneous area ipsilateral to the tumor at week 2, radiation, and further injections of 2141-V11 in the cervical perilymphatic subcutaneous area ipsilateral to the tumor.
  Interventions: Drug: D2C7-IT; Drug: 2141-V11

INTERVENTIONS:
Drug: D2C7-IT — D2C7-IT will be dosed at 166,075 ng in 36 mL.
Drug: 2141-V11 — 2141-V11 will be dosed at 3 mg in 3.5 mL for CED administration. 2141-V11 in the cervical perilymphatic subcutaneous area will be dosed at 2 mg.

SUMMARY:
The purpose of this research study is to determine the safety and efficacy of administering a single intracerebral (within the brain) dose of investigational compounds called D2C7-immunotoxin (IT) and 2141-V11 in residual disease (within tumor margins) after surgery, followed by later repeated injections of 2141-V11 in the subcutaneous area (under the skin) around the lymph nodes of the head and neck for adults newly diagnosed with a type of cancerous brain tumor called glioblastoma. The word "investigational" means the study drugs are still being tested in research studies and are not approved by the U.S. Food and Drug Administration (FDA).

DETAILED DESCRIPTION:
Within this study, approximately 50 study participants will receive a single infusion of D2C7-IT in the hospital, which is delivered to the tumor margins over 3 days through a catheter placed in the brain, followed by a single infusion of 2141-V11 delivered over 7 hours to the tumor margins through the same catheter. About 2 weeks after intratumoral infusion of D2C7-IT and 2141-V11, participants will have their first subcutaneous (under the skin) injection of 2141-V11 in the area around the lymph nodes of the head and neck on the same side as the tumor. About a week after this injection, participants will start standard radiation therapy (RT), which typically lasts either 3 weeks or 6 weeks depending upon age. Once RT is finished, participants will resume injections in the area around the lymph nodes of the head and neck on the same side as the tumor of 2141-V11 about 1 week later. They will have another injection about 3 weeks after finishing RT and then start a schedule of injections about every 3 weeks for up to a year.

There are risks to the study drugs that are described in this document. Some common risks related to D2C7-IT include: effects related to tumor cells dying (tumor necrosis), effects on normal brain tissue, effects related to catheter placement and removal, effects related to fluid infusion into the brain (intracerebral infusion), and reactions to the D2C7-IT being directly infused in your brain. Risks of 2141-V11 being directly infused in your brain and injected in the area around the lymph nodes of the head and neck could include: cytokine release syndrome (release of immune system cells called cytokines that can cause fever, chills, headache, muscle pain, itching, rash, chest tightness, palpitations, shortness of breath, low blood pressure, nausea, vomiting), swelling and redness in the neck area, overstimulation of your immune system such that it attacks other tissues in your body, elevated liver enzymes, and low platelets in the blood.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years of age at the time of entry into the study
2. Newly diagnosed supratentorial GBM, WHO grade 4, IDH wildtype, MGMT unmethylated (high grade glioma with molecular features of GBM will be eligible under WHO 4 malignant glioma) with residual radiographic non-contrast enhancing disease on the post-2 cycles of adjuvant TMZ MRI amenable to catheter placement. The residual radiographic contrast enhancing disease is ≤ 3 cm in maximal diameter in any plane.
3. Patient must have completed standard of care radiation therapy (typically 59.4-60 Gy over approximately 6 weeks duration if under 65 years old and a minimum of 40 Gy over 3 weeks duration if 65 years or older) in combination with TMZ and 2 cycles of post-radiation, adjuvant TMZ. For patients known to be MGMT promoter unmethylated prior to start of radiation therapy, patients are not mandated to have received TMZ in combination to radiation therapy prior to participating in this trial.
4. Karnofsky Performance Score (KPS) > 70%
5. Able to undergo brain MRI wiht and without contrast
6. Hemoglobin ≥ 9 g/dl prior to catheter placement
7. Platelet count ≥ 100,000/µL unsupported. Because of risks of intracranial hemorrhage with catheter placement, platelet count ≥ 125,000/µl is required for the patient to undergo biopsy and catheter insertion, which can be attained with the help of platelet transfusion
8. Neutrophil count ≥ 1000 prior to catheter placement
9. Creatinine ≤ 1.5 x normal range prior to catheter placement
10. Total bilirubin ≤ 1.5 x upper limit of normal (ULN) prior to catheter placement (Exception: Participant has known or suspected Gilbert's Syndrome for which additional lab testing of direct and/or indirect bilirubin supports this diagnosis. In these instances, a total bilirubin of ≤ 3.0 x ULN is acceptable.)
11. AST/ALT ≤ 2.5 x ULN
12. PT and PTT ≤ 1.2 x normal prior to biopsy. Patients with prior history of thrombosis/embolism are allowed to be on anticoagulation, understanding that anticoagulation will be held in the perioperative period per the neurosurgical team's recommendations. Low molecular weight heparin (LMWH) is preferred. If a patient is on warfarin, the international normalized ratio (INR) is to be obtained and value should be below 2.0 prior to biopsy.
13. Patient or partner(s) meets one of the following criteria:

    1. Non-childbearing potential (i.e. not sexually active, physiologically incapable of becoming pregnant, including any person who is post-menopausal or surgically sterile, or any person who has had a vasectomy). Surgically sterile people are defined as those with a documented hysterectomy and/or bilateral oophorectomy or tubal ligation. Postmenopausal for purposes of this study is defined as 1 year without menses.; or
    2. Childbearing potential and agrees to use one of the following methods of birth control: approved hormonal contraceptives (e.g. birth control pills, patches, implants, or infusions), an intrauterine device, or a barrier method of contraception (e.g. a condom or diaphragm) used with spermicide
14. A signed ICF approved by the IRB will be required for patient enrollment into the study. Patients must be able to read and understand the informed consent document and must sign the informed consent indicating that they are aware of the investigational nature of this study

Exclusion Criteria:

1. Patients who are pregnant or breast-feeding/chestfeeding
2. Patients with an impending, life-threatening cerebral herniation syndrome, based on the assessment of the study neurosurgeons or their designate
3. Patients with severe, active comorbidity, defined as follows:

   1. Patients with an active infection requiring intravenous treatment or having an unexplained febrile illness (Tmax > 99.5°F/37.5°C)
   2. Patients with known immunosuppressive disease or known human immunodeficiency virus infection
   3. Patients with unstable or severe medical conditions such as severe heart disease (New York Heart Association Class 3 or 4)
   4. Patients with known lung (forced expiratory volume in the first second of expiration (FEV1) < 50%) disease
   5. Patients with uncontrolled diabetes mellitus
   6. Patients with albumin allergy
   7. Patients with known HIV or Hepatitis C positive status
   8. Major medical illnesses or psychiatric impairments that, in the investigator's opinion, will prevent administration or completion of protocol therapy
4. Patients who previously received other therapeutic interventions for newly diagnosed GBM with the exception of surgical resection and standard of care concomitant radiation therapy and TMZ and 2 cycles of post-radiation, adjuvant TMZ for their brain tumor
5. Patients who have received concomitant radiation therapy and TMZ ≤ 11 weeks prior to start of D2C7-IT CED infusion
6. Patients with evidence of tumor in the brainstem, cerebellum, or spinal cord, radiological evidence of (actively growing) multifocal disease, tumor crossing the midline, extensive subependymal disease, or leptomeningeal disease
7. Patients on greater than 4 mg per day of dexamethasone within the 2 weeks prior to the start of D2C7-IT infusion
8. Patients with worsening steroid myopathy (history of gradual progression of bilateral proximal muscle weakness, and atrophy of proximal muscle groups)
9. Patients with prior, unrelated malignancy requiring current active treatment with the exception of cervical carcinoma in situ and adequately treated basal cell or squamous cell carcinoma of the skin
10. Patients with active autoimmune disease requiring systemic immunomodulatory treatment within the past 3 months
11. Patients who cannot undergo MRI due to obesity or to having certain metal in their bodies (i.e. pacemakers, infusion pumps, metal aneurysm clips, metal prostheses, joints, rods, or plates) or patients with any known severe allergies to contrast agents. Patients with mild allergies (i.e., rash only) are allowed to enroll and will be pretreated with acetaminophen and diphenhydramine prior to injection of the contrast agent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2023-09-06 (Actual); Primary Completion 2026-10-31 (Estimated); Study Completion 2028-10-31 (Estimated)

PRIMARY OUTCOMES:
Median survival defined as the time between initiation of treatment with D2C7-IT in combination with 2141-V11 and death, or last follow up if alive. | 3 years

SECONDARY OUTCOMES:
Safety as measured by the proportion of patients with unacceptable adverse events due to the combination of D2C7-IT and 2141-V11 administered via CED | 6 months
Safety as measured by the proportion of patients with unacceptable adverse events due to pre-radiation therapy administration of cervical perilymphatic injections of 2141-V11, or delayed completion of radiation therapy | 6 months
Safety as measured by 6-month progression-free survival (PFS6) | 6 months
Median PFS will be reported, which is defined as the median time between initiation of D2C7-IT and 2141-V11 infusion treatment and initial failure (disease progression or death). | 18 months

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Landi, MD, Principal Investigator — Duke University
Locations (1):
- Duke University Medical Center, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: The Preston Robert Tisch Brain Tumor Center — https://tischbraintumorcenter.duke.edu/
- See also: Duke Health — https://www.dukehealth.org/clinical-trials